CLINICAL TRIAL: NCT03593603
Title: An Evaluation of Plethysmography-based Trending of Respiratory Rate Using the Nellcor™ Bedside Respiratory Patient Monitoring System
Brief Title: Trending of Respiratory Rate Using the Nellcor™ Bedside Respiratory Patient Monitoring System
Acronym: RespRate
Status: Completed | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: MDT17002NELLRR
Record Dates: First submitted 2018-07-10; First posted 2018-07-20 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Patients Prescribed Non-invasive Respiratory Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Nellcor™ Bedside Respiratory Monitoring System: Patients on the general care floor who are prescribed non-invasive respiratory monitoring via spot check vital signs at least every 4 hours
  Interventions: Device: Nellcor™ Bedside Respiratory Monitoring System

INTERVENTIONS:
Device: Nellcor™ Bedside Respiratory Monitoring System — Nellcor™ Bedside Respiratory Patient Monitoring System with Nellcor™ Respiration Rate Software and the Nellcor™ Adult Respiratory Sensor to provide continuous respiration rate monitoring

SUMMARY:
This is an open-label, non-randomized, prospective, descriptive study of the Nellcor™ Bedside Respiratory Patient Monitoring System using the Nellcor™ Respiration Rate parameter and Nellcor™ Adult Respiratory Sensor The study is intended to gain further information in the clinical space on the function of the Nellcor™ Respiration Rate parameter. The primary objective is to describe spot check (e.g. manual observation) of respiration rate versus cumulative automated counting (trend) of respiratory rate as measured using the Nellcor™ Bedside Respiratory Patient Monitoring System with the Nellcor™ Respiration Rate parameter.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older.
2. A patient who meets the weight requirement for the sensor (e.g. >30kg).
3. A patient at the study site on a General Care Floor (surgical or medical/non-surgical to be distributed equally) and prescribed standard vital sign checks.
4. Patient is willing and able to provide written informed consent.

Exclusion Criteria:

1. Expected length of stay is < 4 hours.
2. Patient is pregnant or lactating.
3. Patient has severe contact allergies that may cause a reaction to standard adhesive materials found in pulse oximetry sensors, ECG electrodes, respiration monitor electrodes or other medical sensors.
4. Patient has an abnormality that may prevent proper application of the device.
5. Patient is in atrial fibrillation.
6. Patient has a documented history of frequent premature atrial contractions (PACs) or premature ventricular contractions (PVCs), defined as greater than 3 in 30 seconds or greater than 6 in 60 seconds within the past 3 months.
7. Patient has an implanted pacemaker.
8. Patient has excessive nail polish that cannot be removed or other dye or discoloration of the finger.
9. Patient has diagnosed central apnea or diagnosed significant obstructive sleep apnea.
10. Patient is currently using continuous positive airway pressure (CPAP).
11. Patient is unwilling or unable to sign informed consent.
12. Evidence that the patient cannot understand the purpose and risks of the study and would require a legally authorized representative to sign informed consent.
13. Patient is participating in another potentially confounding clinical study.
14. Extreme motion conditions such as patient is prescribed to walk more than once per hour or is prescribed a medical device resulting in constant movement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be included who provide informed consent, who are prescribed non-invasive respiratory monitoring via spot check vital signs at least every 4 hours and are without any contact skin allergies to adhesives found in standard pulse oximetry sensors. Potential subjects are those who will be admitted to the General Care Floor. The subject pool will be approximately divided equally between medical/non-surgical and surgical patients.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2018-07-11 (Actual); Primary Completion 2019-05-03 (Actual); Study Completion 2019-05-03 (Actual)

PRIMARY OUTCOMES:
Agreement of RR measured by spot checks vs continuous monitoring | at least 4 hours
  Bias and a range of agreement of the differences between RR measured by spot checks and RR measured using the Nellcor™ Bedside Respiratory Patient Monitoring System

CONTACTS AND LOCATIONS:
Overall Officials: Paul J Amoroso, MD, Principal Investigator — MultiCare Institute for Research and Innovation
Locations (2):
- United States (2):
  - St. John Health System, Tulsa, Oklahoma
  - MultiCare Institute for Research & Innovation, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No